CLINICAL TRIAL: NCT06177756
Title: Targeted Approach to Prevent Early Obesity
Acronym: TAPEObesity
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Principal Investigator, Anita Morandi, Professor, Azienda Ospedaliera Universitaria Integrata Verona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TAPE Obesity
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Obesity, Pediatric
Keywords: Obesity; Pediatric; Prevention; Nutrition
MeSH Terms: conditions — Pediatric Obesity; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental)
  Interventions: Behavioral: Nutritional and lifestyle counseling
- Comparator Arm (No Intervention)

INTERVENTIONS:
Behavioral: Nutritional and lifestyle counseling — At risk children Intervention Arm: schedule at least four visits/year with anthropometric monitoring, educate parents on the appropriate diet, active lifestyle from the first year of life, regular self-monitoring of their child's anthropometry and appropriate dietary composition and portion control, provide tailor-made nutritional suggestions.
  Not-at-risk children Intervention Arm: educational website with interactive tools for growth self-monitoring and diverse lifestyle suggestions.
  Arms: Intervention Arm

SUMMARY:
Lead: UNIVR, Partners involved: UNIME, CHU Lille, INSERM-Lille

This is a multi-center (UNIVR, UNIME, CHU Lille) randomized controlled trial aiming at evaluating the effect of a selective intervention directed to parents of newborns. 1500 subjects will be recruited in both arms and evaluated with the "Childhood Obesity Risk Score" (COBRISC), thanks to anamnestic/clinical evaluations and molecular profiling (polygenic risk score) made at the child's birth. Participants of the intervention arm at the top tertile (33%) of the COBRISC, will access an intensive follow-up program (four visits/year on average, with anthropometric monitoring) at the local Obesity Tertiary Center. This will include educating parents on the appropriate diet, active lifestyle from the first year of life, regular self-monitoring of their child's anthropometry, appropriate dietary composition and portion control, as well as tailor-made nutritional suggestions. To ensure a patient-centred approach, the parents participating in the intensive follow-up program will annually give their feedback and suggestions by an anonymous online survey, whose results will be used to adapt interventions according to parents' requests, as possible and appropriate. The children of the intervention arm classified as not-at-risk will benefit from a "soft" intervention, consisting in the access to an educational website specially implemented with interactive tools for growth self-monitoring and diverse lifestyle suggestions. The children of the whole comparator arm will benefit from routine well visits from their general practitioner/paediatrician.

This is based on the following rationale that: (i) targeted approaches imply higher motivation and commitment for parents, more intense care for families and more effectiveness and cost-effectiveness, compared to traditional population-based interventions; and (ii) early preventive trials have not demonstrated durable effects after the end of the intervention (no cascade effect), while uninterrupted intervention and follow-up from infancy to late childhood have proved long lasting results.

The following end-points will be evaluated: Primary: overall percentage of children growing on an obesity trajectory at three years of age in the intervention compared to the comparator arm. Secondary: percentage of children growing on an obesity trajectory at three years of age in the at-risk group of the intervention arm compared to the at-risk group of the comparator arm; physical activity and sedentary behavior at 1.5 years of age (EY-PAQ questionnaire), responsive feeding (Infant Feeding Styles Questionnaire (IFSQ) at 1.5 years of age, and dietary composition at three years of age (dietary diary and food frequency questionnaire) in the at-risk group of the intervention arm compared to the at-risk group of the comparator arm. All the children will be measured at the tertiary centre, at one, two and three years of age, and afterwards at six and ten years of age.

All the intervention components will comply with the ESPGHAN Guidelines about infant feeding and complementary feeding, the Italian Consensus on Prevention and Treatment of Childhood Obesity, the Italian Reference Levels of Assumption of Nutrients and Energy, and the French Ministerial Recommendations about Nutrition and Physical Activity for infants and children.

Who does what: UNIVR will be in charge of the study protocol writing. UNIVR will also provide Italian and French centers with educational and monitoring materials, including the web-based tool for parents. UNIVR will provide monitoring to all centers and will be in charge of deliverables, data analyses, and results publication. INSERM-Lille will perform DNA microarrays and risk assessments in all recruited newborns.

ELIGIBILITY:
Inclusion Criteria:

* New-borns
* Parent/Guardian's informed consent

Exclusion Criteria:

* Severe prematurity or congenital disease or anomaly or perinatal complication likely to imply long-term consequences on the child possibility to be fed and to grow physiologically (COBRISC is intended to be used to predict childhood obesity in healthy infants and the TAPE-Obesity trial does not provide specific programmes for children with impaired capacity to thrive physiologically)
* Family unavailability to plan a regular follow-up at the local Paediatric Obesity Centre

Max Age: 5 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3000 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Overall percentage of children growing on an obesity trajectory at three years of age in the intervention compared to the comparator arm | 3 years

SECONDARY OUTCOMES:
Percentage of children growing on an obesity trajectory at three years of age in the at-risk group of the intervention arm compared to the at-risk group of the comparator arm. | 3 years
Physical activity and sedentary behavior at 1.5 years of age (EY-PAQ questionnaire) in the at-risk group of the intervention arm compared to the at-risk group of the comparator arm. | 1.5 years
Responsive feeding (Infant Feeding Styles Questionnaire (IFSQ) at 1.5 years of age in the at-risk group of the intervention arm compared to the at-risk group of the comparator arm. | 1.5 years
Dietary composition at three years of age (dietary diary and food frequency questionnaire) in the at-risk group of the intervention arm compared to the at-risk group of the comparator arm. | 3 years

IPD SHARING:
Plan to Share IPD: No